CLINICAL TRIAL: NCT04000165
Title: A Pilot Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Escalating Multiple Oral Doses of AG-348 in Subjects With Stable Sickle Cell Disease
Brief Title: A Dose-Finding Study of AG-348 in Sickle Cell Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Swee Lay Thein, M.D., Swee Lay Thein, M.D., National Institutes of Health Clinical Center (CC)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 190097; 19-H-0097
Record Dates: First submitted 2019-06-22; First posted 2019-06-27 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Sickle Cell Disease
Keywords: HbS polymerization; pyruvate kinase; 2,3- diphosphoglycerate; ATP in red blood cells; acute sickle pain
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — mitapivat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-348 in participants with Sickle Cell Disease (Experimental): Intra-patient dose escalating study, starting with 5 mg twice a day, increasing to 20 mg twice a day, to maximum 50 mg or 100 mg twice a day. Dosing period is every 2 weeks at each dose level. Dose taper will start on Day 42 (50 mg) or Day 56 (100 mg) with dose reduced over 12 to 15 days.
  Interventions: Drug: AG-348

INTERVENTIONS:
Drug: AG-348 — This is a nonrandomized, intra-patient dose escalating clinical study. AG-348 will be administered starting at 5 mg twice a day, increasing to 20 mg twice a day, to maximum 50 mg or 100 mg twice a day. Dosing period is every 2 weeks at each dose level. Dose taper will start on Day 42 (50 mg) or Day 56 (100 mg) with dose reduced over 12 to 15 days.
  Other Names: Mitapivat

SUMMARY:
Background:

Sickle Cell Disease (SCD) is an inherited blood disorder. People with SCD have abnormal hemoglobin in their red blood cells. Researchers are investigating the safety and efficacy of an investigational medicine called AG-348 (mitapivat sulfate) to determine if it will help people with SCD.

Objective:

To test the tolerability and safety of AG-348 in people with SCD.

Eligibility:

People ages 18 and older with SCD.

Design:

Participants will have 8 visits over approximately 14 weeks. At the first visit participants will be screened with a medical history, a physical exam, blood and urine testing, and an EKG. During the following 5 visits, participants will stay at the clinic for 1 night each. Participants will take study drug in increasing doses up to visit 6, after which the drug will be tapered off. All visits will include physical exam, blood, and urine tests. The last visit will occur 4 weeks after stopping the drug. Participants will provide DNA from the blood samples they provide. The DNA will be tested for an inherited gene that can cause differences in response to the study drug. Researchers may also test other genes to see if they can find any genes that interact with SCD.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a multisystem disorder associated with episodes of acute clinical events and progressive organ damage. Episodic pain, triggered by micro-vasoocclusion induced by sickled red blood cells, is the most common acute complication and the leading cause of hospitalization. Management strategies for SCD have evolved very slowly, and treatment of acute pain is still limited to supportive therapy with opioid medication. Until recently in 2017, the only approved therapy for SCD was hydroxyurea (HU), indicated to reduce frequency of acute painful crises but not universally effective. In addition to HU, transfusions with normal red blood cells are widely used to treat severe sickle crises, but this strategy has limitations (not uniformly accessible, accompanied by risks of alloimmunization, hemolytic transfusion reactions and transfusional iron overload). The only curative treatment is bone marrow transplantation, but this option carries significant risks and is limited by the availability of histocompatible donors.

As the root cause of SCD is polymerization of deoxy-HbS, there is a strong rationale for exploring agents that could inhibit/ reduce the polymerization process itself. HbS polymerizes only when deoxygenated, its oxygenation is influenced by a few factors, one key factor being the 2,3- diphosphoglycerate (2,3-DPG) concentration in the red blood cell. 2,3-DPG decreases oxygen binding by preferentially binding to the low oxygen-affinity T conformation of HbS and also stabilizes the T form of hemoglobin S and HbS fiber. In addition, increased 2,3- DPG concentration decreases intracellular red cell pH further promoting HbS polymerization. 2,3-DPG is an intermediate substrate in the glycolytic pathway, the only source of ATP production in red blood cells. Pyruvate kinase (PK) is a key enzyme in the final step of glycolysis; PK converts phosphoenolpyruvate to pyruvate, creating 50% of the total red cell ATP that is essential for maintaining integrity of the red cell membrane. Reduced PK activity leads to accumulation of the upstream enzyme substrates, including 2,3- DPG, that favors polymerization of deoxy-HbS. In humans with SCD, and even in sickle carriers who are generally asymptomatic, reduced oxygen affinity will favor deoxygenation of HbS and its polymerization, and thus sickling. Indeed, the combination of PK deficiency and sickle cell trait causing an acute sickling syndrome has been previously reported in two cases.

Current approaches to reduce HbS polymerization include fetal hemoglobin induction via multiple strategies and drugs that targets HbS polymerization through increasing affinity of hemoglobin for oxygen (eg. Oxbryta (TM) / Voxelotor / GBT440).

Increasing red cell PK (PK-R) activity, leading to a decrease in intracellular 2,3-DPG concentration, presents a potentially attractive therapeutic target for thwarting HbS polymerization and acute sickle pain. AG-348 / mitapivat is a novel, orally bioavailable, small molecule allosteric activator of PK-R, that is currently in Phase II/III clinical trials in humans with PK deficiency (NCT02476916, NCT03548220 / AG348-C-006; NCT03559699 / AG348-C-007). Overview of the preclinical AG-348 data and other data support dose-dependent changes in blood glycolytic intermediates consistent with glycolytic pathway activation at all multiple ascending doses tested, supporting the potential role of AG-348 in the treatment of sickle cell disease. The overall objective of the present study is to determine the clinical safety and tolerability of AG-348 in subjects with SCD.

ELIGIBILITY:
* INCLUSION CRITIERIA:

For enrollment, subjects must meet all of the following criteria during the screening period:

1. Have provided signed written informed consent prior to performing any study procedure, including screening procedures.
2. Age between 18-70 years
3. Unequivocal diagnosis of HbSS confirmed by hemoglobin electrophoresis performed on patients at least 90 days after a blood transfusion if previously transfused, or DNA genotyping
4. No transfusion in the 90 days prior to the first dose of study drug or absence of HbA on hemoglobin analysis (by high-performance liquid chromatography; HPLC)
5. Have adequate organ function, as defined by:

   1. Serum aspartate aminotransferase (AST) less than or equal to 2.5 (SqrRoot) Upper Limit of Normal (ULN) (unless the increased AST is assessed by the Investigator as due to hemolysis and/or hepatic iron deposition) and alanine aminotransferase (ALT) less than or equal to 2.5 (SqrRoot) ULN (unless the increased ALT is assessed by the Investigator as due to hepatic iron deposition).
   2. Serum creatinine less than or equal to 1.25 (SqrRoot) ULN. If serum creatinine is >1.25 (SqrRoot) ULN, then glomerular filtration rate (based on creatinine) must be greater than or equal to 60 mL/min.
   3. Absolute neutrophil count greater than or equal to 1.0 (SqrRoot) 10^9/L.
   4. Hemoglobin greater than or equal to 7 g/dL
   5. Platelet count greater than or equal to 100 (SqrRoot) 10^9/L.
   6. Activated partial thromboplastin time and international normalized ratio less than or equal to 1.5 (SqrRoot) ULN, unless the subject is receiving therapeutic anticoagulants.
6. For women of reproductive potential, have a negative serum or urine pregnancy test during the screening period. Women of reproductive potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy, or tubal occlusion; or who have not been naturally postmenopausal (i.e., who have not menstruated at all for at least the preceding 12 months prior to signing informed consent and have an elevated follicle-stimulating hormone level indicative of menopause during the screening period).
7. For women of reproductive potential as well as men and their partners who are women of reproductive potential, be abstinent as part of their usual lifestyle, or agree to use 2 effective forms of contraception from the time of giving informed consent, during the study, and for 28 days for women and 90 days for men following the last dose of study treatment. An effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, and barrier methods.
8. Be willing to comply with all study procedures for the duration of the study.

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria during screening will not receive AG348 and will not be counted toward the final enrollment count for statistical purposes:

1. Documented pyruvate kinase deficiency
2. Have a significant medical condition that confers an unacceptable risk to participating in the study, and/or that could confound the interpretation of the study data. Such significant medical conditions include, but are not limited to the following:

   1. Poorly controlled hypertension (defined as systolic blood pressure [BP] >150 mmHg or diastolic BP >90 mmHg) refractory to medical management.
   2. History of recent (within 6 months prior to signing informed consent) congestive heart failure; myocardial infarction or unstable angina pectoris; hemorrhagic, embolic, or thrombotic stroke; deep venous thrombosis; or pulmonary or arterial embolism.
   3. Cardiac dysrhythmias judged as clinically significant by the Investigator.
   4. Heart-rate corrected QT interval-Fredericia's method (QTcF) >480 msec with the exception of subjects with right or left bundle branch block.
   5. Clinically symptomatic cholelithiasis or cholecystitis. Prior cholecystectomy is not exclusionary. Subjects with symptomatic cholelithiasis or cholecystitis may be rescreened once the disorder has been treated and clinical symptoms have resolved.
   6. History of drug-induced cholestatic hepatitis.
   7. Iron overload sufficiently severe to result in a clinical diagnosis by the Investigator of cardiac (e.g., clinically significant impaired left ventricular ejection fraction), hepatic (e.g., fibrosis, cirrhosis), or pancreatic (e.g., diabetes) dysfunction.
   8. Have a diagnosis of any other congenital or acquired blood disorder, or any other hemolytic process as defined by a positive direct antiglobulin test (DAT), except mild allo-immunization as a consequence of transfusion therapy.
   9. Positive test for hepatitis B surface antigen or hepatitis C virus (HCV) antibody (Ab) with signs of active hepatitis B or C virus infection. If the subject is positive for HCV Ab, a reverse transcriptase-polymerase chain reaction test will be conducted. Subjects with hepatitis C may be rescreened after receiving appropriate hepatitis C treatment.
   10. Positive test for human immunodeficiency virus 1 or 2 Ab.
   11. Active infection requiring any use of systemic antimicrobial agents (parenteral or oral) or Grade greater than or equal to 3 in severity (per National Cancer Institute Common Terminology Criteria for Adverse Events) within 2 months prior to signing informed consent.
   12. Diabetes mellitus judged to be under poor control by the Investigator or requiring >3 antidiabetic agents, including insulin (all insulins are considered 1 agent); use of insulin per se is not exclusionary.
   13. History of any primary malignancy, with the exception of: curatively treated nonmelanomatous skin cancer; curatively treated cervical or breast carcinoma in situ; or other primary tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years.
   14. Unstable extramedullary hematopoiesis that could pose a risk of imminent neurologic compromise.
   15. Current or recent history of psychiatric disorder that, in the opinion of the Investigator or Medical Monitor, could compromise the ability of the subject to cooperate with study visits and procedures.
   16. Are currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo. Sickle cell anemia subjects on hydroxyurea or L-glutamine will also be considered, provided that they have been on an unchanged dose of hydroxyurea or L-Glutamine for three months prior to enrollment.
   17. Have exposure to any investigational drug, device, or invasive procedure within 3 months prior to the first dose of study treatment. All noninvestigational invasive procedures within 3 months of starting study treatment may be considered as a potential exclusion criteria per the PI s discretion.
   18. Have had any prior treatment with a pyruvate kinase activator.
   19. Have received crizanlizumab or voxelotor in the 12 weeks prior to signing consent
   20. Have a prior bone marrow or stem cell transplant.
   21. Are currently pregnant or breastfeeding.
   22. Are currently receiving medications that are strong inhibitors of cytochrome P450 (CYP)3A4 or strong inducers of CYP3A4 that have not been stopped for a duration of at least 5 days or a timeframe equivalent to 5 half-lives (whichever is longer) prior to the first dose of AG-348.
   23. Are currently receiving hematopoietic stimulating agents (e.g., erythropoietins, granulocyte colony stimulating factors, thrombopoietins) that have not been stopped for a duration of at least 28 days prior to the first dose of study treatment.
   24. Have a history of allergy to sulfonamides if characterized by acute hemolytic anemia, drug-induced liver injury, anaphylaxis, rash of erythema multiforme type or Stevens-Johnson syndrome, cholestatic hepatitis, or other serious clinical manifestations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant results data will be made available 6 months after publication date for a period of 5 year by sending a request to sweelay.thein@nih.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication date for a period of 5 year

REFERENCES:
- [Derived] Le K, Wang X, Chu J, Lundt M, Lee YY, Conrey A, Frey I, Giannini S, Kosinski PA, Hausman JM, Low PS, Jeffries N, Desai SA, Thein SL. Activating pyruvate kinase improves red blood cell integrity by reducing band 3 tyrosine phosphorylation. Blood Adv. 2024 Nov 12;8(21):5653-5662. doi: 10.1182/bloodadvances.2024013504. PMID 39265169
- [Derived] Xu JZ, Conrey A, Frey I, Gwaabe E, Menapace LA, Tumburu L, Lundt M, Lequang T, Li Q, Glass K, Dunkelberger EB, Iyer V, Mangus H, Kung C, Dang L, Kosinski PA, Hawkins P, Jeffries N, Eaton WA, Lay Thein S. A phase 1 dose escalation study of the pyruvate kinase activator mitapivat (AG-348) in sickle cell disease. Blood. 2022 Nov 10;140(19):2053-2062. doi: 10.1182/blood.2022015403. PMID 35576529
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-H-0097.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the National Institutes of Health in Bethesda, Maryland from July 2019 to June 2021.
Period: Overall Study
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Started | 17
Completed Study at 50 mg Dose | 7
Escalated to 100 mg | 10
Completed | 15
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number Participants With Most Common Reported Drug Related Adverse Events
Description: To assess the clinical safety and tolerability of multiple escalating doses of AG-348, an allosteric activator of the enzyme pyruvate kinase, in subjects with stable sickle cell disease (SCD). Safety and tolerability were assessed by frequency and severity of adverse events (AEs) using Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 17
Participants
  Insomnia | 6
  Arthralgia | 3
  Hypertension | 3

2. Primary Outcome: Number Participants With Serious Adverse Events That Were Possibly Drug-related Serious Adverse Events
Description: as for outcome 1
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 17
Participants | 2

3. Primary Outcome: Number Participants With Increase of ≥ 1 g/dL in Hemoglobin
Description: To assess the clinical safety and tolerability of multiple escalating doses of AG-348, an allosteric activator of the enzyme pyruvate kinase, in subjects with stable sickle cell disease (SCD). Safety and tolerability were assessed by defined as a ≥ 1 g/dL increase in hemoglobin at any dose level compared to baseline.
Time Frame: 14 weeks
Population: One participant, withdrawn 3 days after starting the study for a pre-existing pulmonary embolus, was not evaluable for response. Intention to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
Participants | 9

4. Secondary Outcome: Change in Hemoglobin at Each Dose Level of AG-348
Description: To assess change in hemoglobin in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: One participant, withdrawn 3 days after starting the study for a pre-existing pulmonary embolus, was not evaluable for response. 10 participants escalated to 100 mg dose with 1 participant self-discontinued 3 days after escalating to 100 mg dose. Intention to treat analysis.
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
g/dL
  Baseline | 8.73 (0.51)
  5 mg dose of AG-348 | 0.34 (0.22)
  20 mg dose AG-348 | 0.76 (0.22)
  50 mg dose AG-348 | 1.19 (0.22)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | 0.92 (0.26)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | 0.34 (0.22)
  End of Study AG-348 | 0.37 (0.22)

5. Secondary Outcome: Change in Lactic Acid Dehydrogenase (LDH) at Each Dose Level of AG-348
Description: To assess change in lactic acid dehydrogenase (LDH) in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: U/L
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
U/L
  Baseline | 348.4 (51.21)
  5 mg dose of AG-348 | -7.81 (27.81)
  20 mg dose AG-348 | -39.94 (27.81)
  50 mg dose AG-348 | -25.31 (27.81)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | -37.89 (34.95)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | 20.63 (28.35)
  End of Study AG-348 | 30.72 (28.34)

6. Secondary Outcome: Change in Total Bilirubin at Each Dose Level of AG-348
Description: To assess change in total bilirubin in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
mg/dL
  Baseline | 1.82 (0.28)
  5 mg dose of AG-348 | -0.19 (0.17)
  20 mg dose AG-348 | -0.56 (0.17)
  50 mg dose AG-348 | -0.77 (0.17)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | -0.87 (0.2)
  End Of Taper Dose AG-348: number analyzed (Participants) | 15
  End Of Taper Dose AG-348 | -0.19 (0.17)
  End of Study AG-348 | 0.1 (0.17)

7. Secondary Outcome: Change in Absolute Reticulocyte Count at Each Dose Level of AG-348
Description: To assess change in absolute reticulocyte count in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: K/mcL
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
K/mcL
  Baseline | 196.44 (39.88)
  5 mg dose of AG-348 | -20.97 (13.95)
  20 mg dose AG-348 | -20.72 (13.95)
  50 mg dose AG-348 | -44.99 (13.95)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | -34.1 (16.82)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | -13.77 (14.22)
  End of Study AG-348 | 8.1 (14.22)

8. Secondary Outcome: Change in Aspartate Aminotransferase (AST) at Each Dose Level of AG-348
Description: To assess change in aspartate aminotransferase (AST) in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: U/L
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
U/L
  Baseline | 33.88 (5.94)
  5 mg dose of AG-348 | -3.31 (3.43)
  20 mg dose AG-348 | -3.37 (3.43)
  50 mg dose AG-348 | -2 (3.43)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | -3.54 (4.13)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | -2.49 (3.49)
  End of Study AG-348 | 3.02 (3.49)

9. Secondary Outcome: Change in Mean Corpuscular Volume (MCV) at Each Dose Level of AG-348
Description: To assess change in mean corpuscular volume (MCV) in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: fL
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
fL
  Baseline | 103.32 (7.42)
  5 mg dose of AG-348 | -0.5 (0.8)
  20 mg dose AG-348 | 0.52 (0.8)
  50 mg dose AG-348 | 0.42 (0.8)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | 1.98 (1.01)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | -0.25 (0.84)
  End of Study AG-348 | -0.64 (0.82)

10. Secondary Outcome: Change in Fetal Hemoglobin at Each Dose Level of AG-348
Description: To assess the change in fetal hemoglobin (HbF) in stable sickle cell disease participants at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Percent HbF
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
Percent HbF
  Baseline | 20.39 (4.26)
  5 mg dose of AG-348 | -0.42 (0.49)
  20 mg dose AG-348 | -1.02 (0.49)
  50 mg dose AG-348 | -1.31 (0.49)
  100 mg dose AG-348: number analyzed (Participants) | 9
  100 mg dose AG-348 | -0.34 (0.56)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | 0.19 (0.47)
  End of Study AG-348 | 0.81 (0.47)

11. Secondary Outcome: Percent Change From Baseline of 2,3-DPG at Each Dose Level of AG-348
Description: To understand the mechanisms of action of AG- 348 on the glycolytic pathway in sickle cell disease through laboratory studies of specific pharmacodynamics of 2,3-DPG at each dose level of AG-348.
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
percent change
  5 mg Dose AG-348 | -3.74 (3.65)
  20 mg Dose AG-348 | -16.08 (3.65)
  50 mg Dose AG-348 | -23.49 (3.65)
  100 mg Dose AG-348: number analyzed (Participants) | 9
  100 mg Dose AG-348 | -24.13 (4.12)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | 1.97 (3.68)
  End of Study AG-348 | 9.11 (3.68)

12. Secondary Outcome: Percent Change From Baseline of Adenosine Triphosphate (ATP) at Each Dose Level of AG-348
Description: To understand the mechanisms of action of AG- 348 on the glycolytic pathway in sickle cell disease through laboratory studies of specific pharmacodynamics of adenosine triphosphate (ATP) at each dose level of AG-348.
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
percent change
  5 mg Dose AG-348 | 13.68 (6.29)
  20 mg Dose AG-348 | 26.95 (6.29)
  50 mg Dose AG-348 | 33.43 (6.29)
  100 mg Dose AG-348: number analyzed (Participants) | 9
  100 mg Dose AG-348 | 39.84 (6.74)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | 15.51 (6.31)
  End of Study AG-348 | 12.03 (6.31)

13. Secondary Outcome: Percent Change From Baseline in Oxygen Binding p50 Value at Each Dose Level of AG-348
Description: Measure percent change from baseline in oxygen binding p50 value at each dose level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
Percent Change
  5 mg Dose AG-348 | 0.5 (2.88)
  20 mg Dose AG-348 | -2.09 (3.01)
  50 mg Dose AG-348 | -3.84 (3.19)
  100 mg Dose AG-348: number analyzed (Participants) | 9
  100 mg Dose AG-348 | -4.88 (3.9)
  End of Taper Dose AG-348: number analyzed (Participants) | 15
  End of Taper Dose AG-348 | 7.97 (3.1)
  End of Study AG-348 | 10.79 (3.39)

14. Secondary Outcome: Percent Change in Time (Mins) at Which 50% of Red Blood Cells Are Sickled (t50) Value at Each Dose Level of AG-348
Description: Measure percent change in Time (mins) at which 50% of red blood cells are sickled (t50) Value at Each Dose Level of AG-348
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
percent change
  5 mg Dose AG-348 | -0.46 (9.68)
  20 mg Dose AG-348 | 10.19 (9.75)
  50 mg Dose AG-348 | 7.11 (9.84)
  100 mg Dose AG-348: number analyzed (Participants) | 9
  100 mg Dose AG-348 | 13.98 (12.44)
  End of Taper AG-348: number analyzed (Participants) | 15
  End of Taper AG-348 | -11.38 (9.76)
  End of Study AG-348 | 1.67 (10.13)

15. Secondary Outcome: Percent Change of PK-R at Each Dose Level of AG-348
Description: To understand the mechanisms of action of AG- 348 on the glycolytic pathway in sickle cell disease through laboratory studies of specific pharmacodynamics of PK-R at each dose level of AG-348.
Time Frame: 14 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | AG-348 in Participants With Sickle Cell Disease
Number analyzed (Participants) | 16
percent change
  5 mg Dose AG-348 | -6.89 (6.94)
  20 mg Dose AG-348 | -2.82 (6.94)
  50 mg Dose AG-348 | -10.66 (6.94)
  100 mg Dose AG-348: number analyzed (Participants) | 9
  100 mg Dose AG-348 | -28.99 (7.7)
  End of Taper AG-348: number analyzed (Participants) | 15
  End of Taper AG-348 | -8.38 (6.98)
  End of Study AG-348 | -16.47 (6.98)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All Adverse Events (serious and non-serious) spontaneously reported by the subject and/or in response to an open question from study personnel or revealed by observation, physical examination, or other diagnostic procedures will be recorded. AE were pre-specified to be collected as a single Arm/Group irrespective of dose level.
Groups:
- AG-348 in Participants With Sickle Cell Disease: Intra-patient dose escalating, starting with 5 mg twice a day, increasing to 20 mg twice a day, to maximum 50 mg or 100 mg twice a day. Dosing period is every 2 weeks at each dose level. Dose taper will start on Day 42 (50 mg) or Day 56 (100 mg) with dose reduced over 12 to 15 days.
Arm/Group | AG-348 in Participants With Sickle Cell Disease
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG-348 in Participants With Sickle Cell Disease (N=17)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 4 (4)
Pain (General disorders) | 1 (1)
Thromboembolic event: Pulmonary embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG-348 in Participants With Sickle Cell Disease (N=17)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Elevated C-Reactive Protein (CRP) (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Corneal scar (Eye disorders) | 1 (1)
Red eye (bilateral) (Eye disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Helicobacter Pylori (Gastrointestinal disorders) | 2 (2)
Vomiting and diarrhea (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (3)
Fever (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Upper respiratory infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Finger laceration (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bicarbonate decreased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (3)
CPK increased (Investigations) | 4 (4)
Creatinine increased (Investigations) | 1 (1)
Blood urea nitrogen increased (Investigations) | 1 (1)
Chloride increased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 3 (3)
Urine urobilinogen increased (Investigations) | 1 (1)
White blood cell increased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 3 (4)
Thromboembolic event: Pulmonary embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04000165/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT04000165/ICF_002.pdf